CLINICAL TRIAL: NCT04895501
Title: Effects of Shoe Longitudinal Bending Stiffness on Changes in Energy Cost of Running During a 21 km Run
Brief Title: Effects of Shoe Longitudinal Bending Stiffness
Acronym: FAT-FLEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 21CH034; 2021-A00726-35 (Other: ANSM)
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Runners
Keywords: NEUROMUSCULAR FATIGUE; ENERGETIC COST OF RUNNING; LONGITUDINAL BENDING STIFFNESS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- running with stiff shoes (Active Comparator): 21 km of running with stiff shoes followed by a time-to-exhaustion run.
  Interventions: Other: running flexible shoes
- running flexible shoes (Experimental): 21 km of running flexible shoes followed by a time-to-exhaustion run.
  Interventions: Other: running flexible shoes

INTERVENTIONS:
Other: running flexible shoes — 21kms of running flexible shoes followed by a time-to-exhaustion run.

SUMMARY:
Carbon plates inserted in competitive running shoes have been increasingly used in the past 2-3 years and several investigations have shown that these plates increase the longitudinal bending stiffness (LBS) of the shoe. It leads to a redistribution of muscle work and to a modification of the force generation conditions, which may reduce the energy cost of running (Cr) and improve performance.

DETAILED DESCRIPTION:
Only one study has investigated the effects of LBS in running bouts longer than 8 minutes but on the biomechanics part, and their effects on neuromuscular fatigue and prolonged running performance. The aim of this study is to compare shoes with and without carbon plates during a prolonged (21 km) running exercise on Cr, plantar flexor neuromuscular fatigue and running kinetics and kinematics to estimate the changes high-LBS may induce on fatigue and subsequent performance.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 18 and ≤ 50 years.
* men
* experienced, well-trained endurance runners with the capacity to run 21km in less than 1h 40 and who train more than 5h a week.
* free from muscular, bone or joint injuries
* free from neurologic disease
* approval received from a physician

Exclusion Criteria:

* currently participating in a structured exercise program
* injury in the 3 months prior to the protocol
* chronic joint pathologies (e.g.: repetitive sprains, patellar or ligament problems)
* the intake of corticosteroids within 3 months (inhalation, infiltration or history of prolonged corticosteroid therapy).

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
energy cost of running | during the last 4 minutes of a 21km race
  amount of energy needed to travel a unit of distance

SECONDARY OUTCOMES:
ankle plantar flexors | during the last 4 minutes of a 21km race
  ankle plantar flexors maximal voluntary contraction

CONTACTS AND LOCATIONS:
Overall Officials: Léonard FEASSON, Phd, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Unités de Myologie et de Médecine du Sport, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No